CLINICAL TRIAL: NCT05538533
Title: A Phase I Study of Hypofractionated Preoperative Radiation for Head and Neck Cancers (HyPR-HN)
Brief Title: Hypofractionated Preoperative Radiation for Head and Neck Cancers (HyPR-HN)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Joseph Zenga, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO44863
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Hypofractionated Preoperative Radiation; Time-to-Event Continuous Reassessment Methodology; TITE-CRM
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will use a time-to-event continual reassessment method (TITE-CRM) for assigning subjects to the radiation therapy dosages.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 46 Gray (Gy) (Experimental): 46 gy of radiation therapy will be administered in 10 fractions.
  Interventions: Radiation: 46 Gy Radiation Therapy
- 40 Gray (Gy) (Experimental): 40 gy of radiation therapy will be administered in 7 fractions.
  Interventions: Radiation: 40 Gy Radiation Therapy
- 35 Gray (Gy) (Experimental): 35 gy of radiation therapy will be administered in 5 fractions.
  Interventions: Radiation: 35 Gy Radiation Therapy

INTERVENTIONS:
Radiation: 46 Gy Radiation Therapy — Dose per fraction of 4.6.
  Arms: 46 Gray (Gy)
Radiation: 40 Gy Radiation Therapy — Dose per fraction 5.7.
  Arms: 40 Gray (Gy)
Radiation: 35 Gy Radiation Therapy — Dose per fraction 7.0.
  Arms: 35 Gray (Gy)

SUMMARY:
This is a phase 1 study to determine the safety of a condensed preoperative radiation regimen (10, 7, or 5 fractions) for the management of head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
All subjects in this study will receive pre-operative hypofractionated radiation therapy, which will be subject to fractionation reduction, that being 10 fractions, 7 fractions, or 5 fractions, as compared to 30 fractions of conventional radiation therapy. All patients will subsequently undergo surgery for resection of remaining disease at the primary site and at-risk nodal basins 6-8 weeks after completion of radiation.

The subjects will receive smaller number of fractions (total visits) but with a higher dose of radiation with each Dose Level. Participants will receive a total radiation dose of 46 Gy in 10 fractions (Dose Level 1), 40 Gy in 7 fractions (Dose Level 2), or 35 Gy in 5 fractions (Dose Level 3), depending on the assigned experimental total fractions. Radiation will be delivered using intensity modulated radiation therapy (IMRT) with a daily cone-beam CT for five days a week, for less than two weeks depending on the assigned dose level at the time of enrollment.

Due to the novelty of translational data and non-dependency on the primary endpoint, presentation and publication in a scientific journal of the translational endpoints may precede publication of the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older with surgically resectable, Human papillomavirus (HPV) -negative squamous cell carcinoma of the head and neck (squamous cell carcinoma of the larynx, hypopharynx, oropharynx, oral cavity, nasal cavity or paranasal sinuses). Resectability will be determined by the treating surgeon. Patients must have locoregionally advanced disease defined by clinical T3-4 staging and/or clinical node positive staging. Patients may also be eligible if they meet one of the following criteria:

   1. Clinical T2N0 disease with perineural invasion identified on a pretreatment biopsy.
   2. Clinical T2N0 disease with lymphovascular space invasion identified on a pretreatment biopsy.
   3. Clinical T2N0 oral cavity cancer with clinical, biopsy, or radiographic depth of invasion of at least 5 mm.
2. Zubrod performance status 0-2.
3. Patients must have the psychological ability and general health that permits completion of the study requirements and required follow-up.
4. Inclusion of COVID-19 positive patients will be based on standard institutional protocol.
5. Female patients must meet one of the following:

   * Postmenopausal for at least one year before the screening visit, OR
   * Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), OR
   * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agrees to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 90 days after the last dose of study agent, AND
   * Agrees to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, postovulation methods] and withdrawal are not acceptable contraception methods).
6. Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:

   * Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
   * Must also adhere to the guidelines of any study-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, postovulation methods] and withdrawal are not acceptable methods of contraception.
7. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Radiographic evidence of extranodal extension.
2. Patients with laryngeal involvement who are candidates for non-surgical laryngeal preservation as deemed by a surgeon and/or radiation oncologist. These patients include, but are not limited to, those with T1-T3 laryngeal cancer who do not have pretreatment tracheostomy and/or feeding tube or those with base of tongue/hypopharyngeal cancers with laryngeal involvement without cartilage invasion or pretreatment tracheostomy and/or feeding tube.
3. HPV-positive squamous cell carcinoma.
4. Prior invasive malignancy within the past three years (except for non-melanomatous skin cancer, and early stage treated prostate cancer).
5. Life expectancy less than 12 months.
6. Zubrod performance status ≥ 3.
7. Patients with prior radiation therapy to the head and neck (Note: Prior external beam radiotherapy is excluded, but iodine-131 is allowed).
8. Prior systemic therapy, including cytotoxic chemotherapy, biologic/targeted therapy, or immune therapy for the study cancer.
9. Body weight ≤ 30 kg.
10. Any of the following severe laboratory abnormalities within 14 days of registration, unless corrected prior to it: sodium < 130 mmol/L or > 155 mmol/L; potassium < 3.5 mmol/L or > 6 mmol/L; fasting glucose < 40 mg/dL or > 400 mg/dL; serum calcium (ionized or adjusted for albumin) < 7 mg/dL or > 12.5 mg/dL; magnesium < 0.9 mg/dL or > 3 mg/dL.
11. Unstable angina and/or congestive heart failure requiring hospitalization within three months prior to step 1 registration.
12. Transmural myocardial infarction within three months prior to step 1 registration.
13. Medical or psychiatric illness which would compromise the patient's ability to tolerate treatment or limit compliance with study requirements.
14. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during treatment and for six months after radiation, this exclusion is necessary because the treatment involved in this study may be significantly teratogenic. Women who are breastfeeding are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with a dose-limiting toxicity related to inoperability. | 8 Weeks
  Inoperability after HyPR-HN, is defined as an inability to proceed to surgery within eight weeks of radiation.
The number of subjects with a dose-limiting toxicity related to perioperative complication rates. | 8 Weeks
  Severe perioperative complication rates, defined as unacceptable toxicity from initiation of treatment until 30 days postoperatively (grade 4/5 toxicity) probably or definitely related to treatment.
The number of subjects with severe delayed toxicity. | Up to one year
  Severe delayed toxicities, defined as any unacceptable toxicity (grade 4+) after 30 days postoperatively until one year after initiation of HyPR-HN probably or definitely related to treatment.

SECONDARY OUTCOMES:
Overall survival | One year
  This measure is the number of subjects alive at one year following the conclusion of scheduled radiation therapy.
Recurrence-free Survival | One year
  This measure is the number of subjects who are survival free of locoregional recurrence or distant metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zenga, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No